CLINICAL TRIAL: NCT04417348
Title: Expression of Opsins Receptors in Melasma and Its Modification With UV-Visible Light Sunscreen and 0.05% Retinoic Acid.
Brief Title: Opsin Receptors in Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Adjunt professor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPN3Mel
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: patients with melasma divided in a UV-Visible light filter with 0.05% retinoic acid group and UV-Visible light filter alone
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinoic Acid (Active Comparator): patients with melasma treated with 0.05% retinoic acid plus UV-Visible light filter
  Interventions: Drug: Retinoic acid
- Sunscreen (Placebo Comparator): patients with melasma treated with UV-Visible light filter alone
  Interventions: Drug: Retinoic acid

INTERVENTIONS:
Drug: Retinoic acid — To evaluate the role of Opsin receptors in melasma. The patients were treated with 0.05% Retinoic Acid, a regular therapy to treatment melasma, a ligand of Opsin receptors. Also, Uv-Visible light filter treatment as a posible opsin receptor blocker

SUMMARY:
Melasma is a hyperpigmentation disorder that is probably exacerbated by visible light. Opsin receptors (OPN 1, 2, 3, 4 y 5) were described in the skin, being capable of activating melanogenesis induced by visible light. The aim of this study was to evaluate the expression of OPN in melasma skin and its changes following treatment with UV-Vis filter and 0.05% retinoic acid for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with melasma, of 18 years of age and older, without previous treatment or photoprotection measures within the previous 4 weeks, who had Melasma Activity and Severity Index (MASI) scores higher than 7

Exclusion Criteria:

* pregnancy or nursing, menopause, coexistence of other pigmentation conditions, heat exposure, regular exercise, diet restriction, consumption of food supplements or any type of drugs (including anti-inflammatories and hormonal treatments) within the previous 2 months, and women who had given birth within 1 year

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
MASI score | 3 months
  Melasma Activity and Severity Index

SECONDARY OUTCOMES:
Opsin receptors | 3 months
  Relative Expression of the opsin receptors by RT-qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Regazzetti C, Sormani L, Debayle D, Bernerd F, Tulic MK, De Donatis GM, Chignon-Sicard B, Rocchi S, Passeron T. Melanocytes Sense Blue Light and Regulate Pigmentation through Opsin-3. J Invest Dermatol. 2018 Jan;138(1):171-178. doi: 10.1016/j.jid.2017.07.833. Epub 2017 Aug 24. PMID 28842328
- [Result] Ozdeslik RN, Olinski LE, Trieu MM, Oprian DD, Oancea E. Human nonvisual opsin 3 regulates pigmentation of epidermal melanocytes through functional interaction with melanocortin 1 receptor. Proc Natl Acad Sci U S A. 2019 Jun 4;116(23):11508-11517. doi: 10.1073/pnas.1902825116. Epub 2019 May 16. PMID 31097585